CLINICAL TRIAL: NCT03157765
Title: A Randomized Study on the Value of an Endometrial Scratch Prior to a Frozen Embryo Transfer Cycle in the Treatment of Recurrent Implantation Failure
Brief Title: Trial of Endometrial Scratch Prior to Frozen Embryo Transfer in Patients With Recurrent Implantation Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research site
Sponsor: Brown Fertility (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB for RIP/FET
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Implantation Failure in Setting of Artifically Prepared Endometrium
Keywords: recurrent implantation failure; frozen embryo transfer; IVF; endometrial scratch; endometrial injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMB intervention (Experimental): These patients receive and endometrial biopsy
  Interventions: Procedure: endometrial biopsy
- Routine care (No Intervention): These patient receive routine care

INTERVENTIONS:
Procedure: endometrial biopsy — endometrial biopsy
  Arms: EMB intervention

SUMMARY:
Patients with a history of recurrent implantation failure who are planning a frozen embryo transfer (FET) are enrolled into the program. Patients are randomized to an endometrial biopsy prior to starting estrogen to prepare for the transfer of warmed vitrified embryos or to routine care.

DETAILED DESCRIPTION:
Patients who failed to achieve a clinical pregnancy after embryo transfer of at least three high quality embryos in at least two IVF or FET cycles and for whom their last failed cycle was a frozen embryo transfer are offered the opportunity to enroll in this study. All patients will follow our routine FET protocol.

On a randomized basis, selected patients will undergo an endometrial biopsy using a Pipelle disposable device in the week prior to starting estrogen to prepare her endometrium.

ELIGIBILITY:
Inclusion Criteria:

* At least two prior consecutive failed IVF or FET cycles with transfer of at least 3 high quality embryos and with last cycle a FET cycle

Exclusion Criteria:

* Alternate explanation for implantation failure (e.g., intrauterine pathology)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | within 6 months after recruitment
  Sacs seen in early ultrasound divided by the number of embryos transferred
clinical pregnancy rate | within 6 months after recruitment
  Number of patients with ultrasound evidence of pregnancy divided by the number of embryo transfers

SECONDARY OUTCOMES:
ongoing pregnancy rate | within 18 months of recruitment
  Viable or delivered pregnancies at conclusion of study divided by the number of embryo transfers
biochemical pregnancy rate | within 6 months after recruitment
  number of positive pregnancy test divided by number of embryo transfers
miscarriage rate | within 18 months after recruitment
  number of losses of clinical pregnancies divided by number of clinical pregnancies